CLINICAL TRIAL: NCT03305185
Title: Efficacy of Scoliosis Specific Exercise (SSE) in Patients With Adolescent Idiopathic Scoliosis (AIS) During Bracing: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Scoliosis Specific Exercise in Patients With Adolescent Idiopathic Scoliosis During Bracing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 16-206
Record Dates: First submitted 2017-09-20; First posted 2017-10-09 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS
MeSH Terms: interventions — Braces

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with AIS referred for bracing through the hospital's specialist outpatient clinic are eligible to enrol the study. The Investigator will document whether each patient meets the selection criteria before enrolment into the study. The Investigator or designee will also obtain an IRB/EC approved Informed consent from each patient and/or guardian.
  Recruited patients will be randomly assigned to either SSE group or control group in a ratio of 1:1. The radiographic evaluation, physical examination and PROM questionnaires will be assessed at baseline, post-treatment 3 months, 6 months, 12 months and until skeletal maturity.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor, statistician and investigator blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth SSE with Bracing (Experimental): Patients in this group will be prescribed an outpatient-based Schroth exercise program, as per our preliminary study. It consists of an individualised eight-week outpatient program that includes four initial private training sessions, once every two weeks, where exercises will be taught to the patient and their caregivers. A home exercise program will be instituted thereafter and patients will be required to return for supervised sessions once every two months.
  Interventions: Combination Product: Schroth SSE with Bracing
- Bracing alone (Active Comparator): Patients in the control group will receive standard level of care for bracing, which consists of education on general exercises for spinal movement, strengthening, and balancing. These patients will only attend study assessments with no extra physiotherapy sessions.
  Interventions: Device: Bracing alone

INTERVENTIONS:
Combination Product: Schroth SSE with Bracing — Patients in this group will be prescribed an outpatient-based Schroth exercise program, as per our preliminary study. It consists of an individualised eight-week outpatient program that includes four initial private training sessions, once every two weeks, where exercises will be taught to the patient and their caregivers. A home exercise program will be instituted thereafter and patients will be required to return for supervised sessions once every two months.
  Arms: Schroth SSE with Bracing
Device: Bracing alone — Patients in the control group will receive standard level of care for bracing, which consists of education on general exercises for spinal movement, strengthening, and balancing. These patients will only attend study assessments with no extra physiotherapy sessions.
  Arms: Bracing alone

SUMMARY:
The purpose of this study is to examine the effectiveness of Schroth scoliosis-specific exercises (SSE) on patients with adolescent idiopathic scoliosis (AIS) during bracing. The goal is to determine if Schroth SSE combined with bracing can is superior in controlling curve progression when compared with bracing alone. Curve progression is defined as worsening of coronal Cobb angle of 6 degrees or more.

DETAILED DESCRIPTION:
Adolescent Idiopathic scoliosis (AIS) is a three-dimensional deformity of the spine, characterized by a lateral curvature and vertebral rotation. Its prevalence is estimated to be 2.5% in children between aged 10 and 16 in Hong Kong. Curve progression occurs during pubertal growth spurt. If the primary curve does not exceed 40 degree at skeletal maturity, it is unlikely to continue to progress, and there are little or no long-term clinical consequences. However, if the curve progresses beyond 50 degree during adolescence, it may cause functional limitation, accelerated disc degeneration with potential neurological deficit, cosmetic concerns, decreased quality of life, and possible progression in adulthood. Thus, surgical correction of the deformity with instrumented spinal fusion is usually recommended if the curve reaches 50 degree during adolescence.

Currently, spinal bracing is the only the only non-operative treatment supported with high-quality evidence that can prevent curve progression. In a randomized controlled trial, Weinstein et al. recently reported in the New England Journal of Medicine that bracing was effective in preventing curve progression to threshold for surgery in 72% of cases. The trial was terminated early due to the treatment benefit in favor of bracing. Nonetheless, the authors reported a treatment failure rate of 25% in the randomized cohort, which was similar to previous published studies. Hence, despite the best available non-operative treatment, the number of adolescents ultimately requiring surgery remains substantial. Surgery is associated with medical comorbidities, can cause psychosocial stress to the children and their families, and has significant financial impact on healthcare, with the total costs of spinal surgery to correct AIS ranked second only to appendicitis among children 10 to 17 years of age. Consequently, further effective strategies to prevent scoliosis progression in children are needed.

Scoliosis-specific exercise (SSE) has been proposed as an additional non-operative intervention that may reduce curve progression during the adolescent growth spurt. However, the standard of care for non-operative treatment of AIS varies widely between North America and Europe, and the use of SSE is not universally accepted. SSE is a potentially low-cost intervention that will be of substantial benefit even if a relative risk reduction in curve progression or reaching the threshold for surgery is reduced in a modest proportion of those participating.

SSE, as opposed to generalized physiotherapy, consists of individually-adapted exercises that aim to promote spinal realignment through self-correction and stabilization, as well as modulating patterns of trunk muscles recruitment. Electromyography (EMG) of paraspinal and abdominal muscles in AIS patients revealed disrupted patterns of muscles recruitment, which are associated with a disparity in trunk isometric rotation strength between sides. AIS patients demonstrate proprioceptive and balance control problems, along with a distorted body schema, resulting in a mismatch between the actual spinal alignment and the patients' internal representation of the body. SSE aims to reverse the anomalous patterns of muscle recruitment through training, and modify the body schema with visual and somatosensory feedback. This forms the theoretical neurophysiological basis for using this treatment strategy for AIS.

Schroth SSE is one of the most studied and widely-used schools of SSE. It is a technique tailored to the type of scoliosis and the curve magnitude of each patient. It is based on vertebrae deflections and sagittal corrections that result in horizontal vertebrae de-rotation. It uses rotational breathing and postural auto-correction to reverse the underlying impairments in spinal muscle function, postural control and proprioception which contribute to the development of curvature in AIS. Patients will also be given cognitive behavioral strategies to empower them to self-manage their conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS
* Male or female from 10 to 15 year-old, inclusive, at the time of consent provided
* Skeletal immaturity, defined as a Risser grade (amount of ossification and eventual fusion of the iliac apophysis) of 0, 1, or 2
* Cobb angle of 25-40
* No prior conservative or surgical treatment for AIS

Exclusion Criteria:

* An underlying cause or association that may cause scoliosis
* Leg length discrepancies or lower limb deformities that may interfere with spinal posture
* Previous spinal surgery
* Cognitive impairment
* Those receiving any other forms of treatment including alternative medicine for the treatment of their scoliosis
* Those who are unable to return for follow-up to complete the trial.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Schroth SSE during bracing versus bracing alone in AIS patients as determined by the difference in coronal Cobb angle pre- and one year post-treatment | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  1. To evaluate the effect of Schroth SSE during bracing versus bracing alone in AIS patients as determined by the difference in coronal Cobb angle pre- and one year post-treatment

SECONDARY OUTCOMES:
Compare changes in sagittal plane radiological parameter between Schroth SSE with bracing and bracing alone by EOS Imaging System | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To evaluate the effect of Schroth SSE during bracing compared with bracing alone on sagittal plane radiological parameter using EOS Imaging System
Compare changes in transverse plane radiological parameter between Schroth SSE with bracing and bracing alone by EOS Imaging System | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To evaluate the effect of Schroth SSE during bracing compared with bracing alone on transverse plane radiological parameter using EOS Imaging System
Compare changes in surface topography between Schroth SSE with bracing and bracing alone using Bunnell's scoliometer | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To evaluate the effect of Schroth SSE during bracing compared with bracing alone on surface topography using Bunnell's scoliometer
Compare changes in surface topography between Schroth SSE with bracing and bracing alone using clinical photography | baseline, 6 months, 12 months, until skeletal maturity
  To evaluate the effect of Schroth SSE during bracing compared with bracing alone on surface topography using clinical photography
Compare changes in surface topography between Schroth SSE with bracing and bracing alone using VITUS Smart XXL 3D body scanner system | baseline, 6 months, 12 months, until skeletal maturity
  To evaluate the effect of Schroth SSE during bracing compared with bracing alone on surface topography using VITUS Smart XXL 3D body scanner system
Measure quality of life between Schroth SSE with underarm brace and underarm brace alone by SRS-7 questionaire | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To measure quality of life between Schroth SSE with underarm brace and underarm brace alone by SRS-7 questionaire
Measure health outcomes between Schroth SSE with underarm brace and underarm brace alone by EQ-5D-5L | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To measure health outcomes between Schroth SSE with underarm brace and underarm brace alone by EQ-5D-5L
Measure patients' perception of their appearance between Schroth SSE with underarm brace and underarm brace alone by Trunk Appearance Perception Scale (TAPS) | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To measure patients' perception of their appearance between Schroth SSE with underarm brace and underarm brace alone by Trunk Appearance Perception Scale (TAPS)
Measure levels of pain between Schroth SSE with underarm brace and underarm brace alone by Numeric Pain Ratings | baseline, 3 months, 6 months, 12 months, until skeletal maturity
  To measure levels of pain between Schroth SSE with underarm brace and underarm brace alone by Numeric Pain Ratings

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh(Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No